CLINICAL TRIAL: NCT01826682
Title: Physiotherapy Program Intervention in Exacerbation of Chronic Obstructive Pulmonary Disease.
Brief Title: Physiotherapy in Exacerbation Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0039UG
Record Dates: First submitted 2013-03-28; First posted 2013-04-08 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, physiotherapy, exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Therapy Modalities; Breathing Exercises; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical treatment (Placebo Comparator): 29 people are being recruited in order to the inclusion criteria for the study. Placebo controlled.
  Interventions: Other: Medical treatment
- Physiotherapy program+medical treatment (Active Comparator): 29 people are recruited in order to the inclusion criteria for the study. Experimental group
  Interventions: Other: Physiotherapy program+medical treatment

INTERVENTIONS:
Other: Physiotherapy program+medical treatment — Patients included in this group are going to receive physiotherapy during their hospital stay 45 minutes every day. The physical training is based on respiratory exercises, the use of a flutter (positive expiratory pressure), pedaling and theraband exercises.
  Other Names: Physiotherapy; Respiratory exercises; Strength exercises
  Arms: Physiotherapy program+medical treatment
Other: Medical treatment — Standard medical treatment without physiotherapy.
  Other Names: Drugs
  Arms: Medical treatment

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic condition. Its evolution can be aggravated in some periods by an increase of the symptoms (above all the cough, the dyspnoea and the quantity of sputum purulence). This is known as exacerbation and it is the most frequent cause of hospital stay, urgences services and death in COPD. A physiotherapy program is carrying out in patients attending to the Hospital because of an exacerbation.

The hypothesis of this study is that a physiotherapy program added to a medical treatment increase the ventilatory function, the physiques variables, decrease depression and anxiety and improve the quality of life. Additionally, it is going to be assessed the effect of physiotherapy in time using phone calls and visits to the patient's home.

DETAILED DESCRIPTION:
The benefits added to the respiratory physiotherapy and physical activity have been evidenced previously in the treatment of COPD. This justify the need of a short physiotherapy intervention program regarding to the hospital stay in exacerbation of COPD and a follow-up after the hospital stay.

4% of europeans have been reported to have medical intervention caused by respiratory exacerbation. 20% of these patients are patients with COPD. The mortality of COPD exacerbation is about 14% and 30% if mechanical ventilation is needed.

In order to that, it is very important to improve the quality of life and the recuperation of patients. It is relevant to mention the the high cost associated to this condition.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with exacerbation.
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion.

Exclusion Criteria:

* Heart disease.
* Neurological patients.
* Contraindications of physiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Strength in upper and lower limbs | baseline, 12 months
  Changes from baseline to postintervention during hospital stay in lower and upper limbs strength. The quadriceps and the hand-grip strength is assessed using a dynamometer with a standard protocol allowing three attempts on each side. During each measurement, patients were sitting with their shoulder adducted and elbow flexed to 90°. The maximum value achieved was used in the analyses. This is important in order to quantify the increase of strength Kg/cm2 The test 2-minute step in place is also going to be used for this purpose, counting the times the patients go up the right knees in two minutes.

SECONDARY OUTCOMES:
Changes in quality of life | baseline, 12 months
  Changes from baseline to postintervention during hospital stay in quality of life associated with health. This is going to be measure with two questionnaires: the EuroQol-5 questionnaire and the Health Questionnaire St. George
Respiratory parameters | baseline, 12 months
  Changes from baseline to postintervention in respiratory parameters using a spirometer as recommended by the American Thoracic Society. The most important respiratory parameters evaluated are forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), carbon dioxide partial pressure (PCO2) and oxygen partial pressure (PO2)
Activity monitoring | baseline
  The accelerometer Armband is going to be used for activity monitoring. It measures the intensity of the activity during 12 hours.
Performance of Physical activity | baseline
  The participants are going to complete the Baecke physical activity questionnaire-modified in order to describe their physical status at baseline.
Changes in quality of sleep | baseline, 12 months
  Changes in quality of sleep from baseline to postintervention. For this purpose, the participants are going to complete the Pittsburgh Quality of Sleep Index. This is a self-rating questionnaire with seven subscores that result in a global score between 0 and 21.
Changes in anxiety and depression | baseline, 12 months
  Changes from baseline to postintervention in anxiety and depression measured with the Hospital Anxiety and Depression Scale. Patients are going to completed this questionnaire composed of statements relevant to either generalised anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PT, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres-Sanchez I, Valenza MC, Cabrera-Martos I, Lopez-Torres I, Benitez-Feliponi A, Conde-Valero A. Effects of an Exercise Intervention in Frail Older Patients with Chronic Obstructive Pulmonary Disease Hospitalized due to an Exacerbation: A Randomized Controlled Trial. COPD. 2017 Feb;14(1):37-42. doi: 10.1080/15412555.2016.1209476. Epub 2016 Aug 11. PMID 27715322
- [Derived] Valenza MC, Valenza-Pena G, Torres-Sanchez I, Gonzalez-Jimenez E, Conde-Valero A, Valenza-Demet G. Effectiveness of controlled breathing techniques on anxiety and depression in hospitalized patients with COPD: a randomized clinical Trial. Respir Care. 2014 Feb;59(2):209-15. doi: 10.4187/respcare.02565. Epub 2013 Jul 23. PMID 23882107